CLINICAL TRIAL: NCT04710420
Title: Prospective Multicenter Registry on the Endovascular Treatment in Critical Limb Threatening Ischemia With Below the Knee Lesions With WIFI Assessment
Brief Title: Prospective Multicenter Registry on the Endovascular Treatment in Critical Limb Threatening Ischemia With Below the Knee Lesions With Wound, Ischemia, and Foot Infection (WIFI) Assessment
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: RenJi Hospital (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); Zhejiang University (Other); First Affiliated Hospital of Zhejiang University (Other); Second Affiliated Hospital of Soochow University (Other); Qingdao Haici Hospital (Other); Chengdu University of Traditional Chinese Medicine (Other); Fudan University (Other); Huashan Hospital (Other)
Responsible Party: Principal Investigator, Lian-Rui Guo, Director, vascular suregry department, Xuanwu Hospital, Beijing
Other Study IDs: PRIME-WIFI
Record Dates: First submitted 2021-01-08; First posted 2021-01-14 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Chronic Limb-threatening Ischemia; Endovascular Therapy
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (4):
- WIfI stage 1: Very low risk of amputation was determined according to the SVS WIfI classification system.
  Interventions: Device: Endovascular therapy
- WIfI stage 2: Low risk of amputation was determined according to the SVS WIfI classification system.
  Interventions: Device: Endovascular therapy
- WIfI stage 3: Moderate risk of amputation was determined according to the SVS WIfI classification system.
  Interventions: Device: Endovascular therapy
- WIfI stage 4: High risk of amputation was determined according to the SVS WIfI classification system.
  Interventions: Device: Endovascular therapy

INTERVENTIONS:
Device: Endovascular therapy — Endovascular treatment for critical limb threatening Ischemia

SUMMARY:
This is a prospective multicenter clinical study that used WIFI grading scores at different periods to evaluate the therapeutic value of endovascular therapy and this grading system for Chronic limb-threatening ischemia.

ELIGIBILITY:
Inclusion Criteria:

1. patients > 18 years of age;
2. patients with Chronic limb-threatening ischemia (CLTI);
3. patients with below-the-knee lesions undergoing endovascular treatment;
4. target limbs with certain WIfI stage;
5. patients voluntary and capable of follow-up;
6. informed consent.

Definition of CLTI:

A diagnosis of CLTI requires objectively documented atherosclerotic PAD in association with ischemic rest pain or tissue loss (ulceration or gangrene).

Exclusion Criteria:

1. Contraindication for antiplatelet , anticoagulant or thrombolytic agent;
2. Contrast agent allergy;
3. Dysfunctional protein C, protein S, antithrombin Ⅲ(AT Ⅲ) or refusal of blood transfusion;
4. Complications affecting surgical safety;
5. Major amputation was adopted to the target extremity;
6. The existence of aneurysm in the target vessels;
7. The existence of perforation, dissection or any other injury requiring intervention in the target vessels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic limb-threatening ischemia.
Sampling Method: Probability Sample
Enrollment: 842 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Freedom from major amputation | 12 months
  Major amputation was defined as any amputation above-the-ankle of the target limb.

SECONDARY OUTCOMES:
WIfI stages | 12 months
  Before follow-up and during each follow-up, the Society for Vascular Surgery wound, ischemia, and foot Infection (WIfI) were evaluated classification system.
Amputation-free survival | 12 months
  Survival without target limb major amputation.
Freedom from all-cause death | 12 months
  Freedom from all-cause death.
Freedom from clinically driven target limb reintervention | 12 months
  Clinically driven target limb reintervention was defined as any reintervention of ipsilateral infrapopliteal arteries for recurrent clinical symptoms.
Freedom from major adverse event | 12 months
  Major adverse event was a composite of major amputation, all-cause death, and clinically driven target limb reintervention.
Quality of life | 12 months
  The Vascular Quality of Life (VascuQol) questionnaire was used to assess QOL score.
Primary sustained clinical improvement | 12 months
  A decrease of at least 1 Rutherford grade without any reintervention.
Hospitalization time | 12 months
  The length of hospital stay was evaluated
Hospitalization expenses | 12 months
  Hospitalization costs for patients were evaluated
Adverse event rates | 1 week
  Adverse event rates includes surgically related arterial dissection, perforation, rupture, embolism, acute thrombosis, pseudoaneurysm and hematoma formation

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China